CLINICAL TRIAL: NCT02416726
Title: Comparison of Gene Mutations Among the Primary Tumor, Matched Metastatic Lymph Node and Peripheral Blood in Advanced Nonsquamous Non-small Cell Lung Cancer Using Next-generation Sequencing
Brief Title: Comparison of Gene Mutations in Matched Samples in Advanced Nonsquamous NSCLC Using NGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Endoscope Department, Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201501
Record Dates: First submitted 2015-03-25; First posted 2015-04-15 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: Gene testing; Next-generation sequecing; Primary tumor; Metastatic lymph node; Peripheral blood
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peripheral blood (Experimental): The peripheral blood sample will be extrated with DNA and performed NGS using Illumina Nextseq500 sequencer.
  Interventions: Device: Nextseq500 sequencer
- Primary tumor (Experimental): The gene testing of the primary tumor tissue diagnosed with nonsquamous NSCLC will be performed with NGS technique using Illumina Nextseq500 sequencer.
  Interventions: Device: Nextseq500 sequencer
- Metastatic lymph node (Experimental): The gene testing of the metastatic lymph node tissue diagnosed with nonsquamous NSCLC will be performed with NGS technique using Illumina Nextseq500 sequencer.
  Interventions: Device: Nextseq500 sequencer

INTERVENTIONS:
Device: Nextseq500 sequencer — The sequencer will be used to detect the gene mutations of the primary tumor, metastatic LN and peripheral blood samples obtained from patients.

SUMMARY:
The objective of the study was to compare the gene mutation status among the primary tumor, matched metastatic lymph node (LN) and peripheral blood in advanced nonsquamous non-small cell lung cancer (NSCLC) using next-generation sequencing (NGS).

DETAILED DESCRIPTION:
Many gene mutations have been detected in lung cancer, which might differ between the primary tumor and the metastases in a same patient. One may cause by the heterogenicity of the tumor, another may cause by the sensitivity of the detection technique. So we determine to use NGS, which is a more sensitive technique, to detect the different gene mutations among the primary tumor, metastatic LN and peripheral blood in advanced nonsquamous NSCLC.

The study was designed as a prospective and single center study. Thirty five patients will be enrolled into the study and the clinical data of the patients, including his smoke history, cancer history, occupation exposure and so on, will be collected and recorded in a case report form. For the patients recruited in the study, the primary tumor and metastatic lymph nodes will be obtained by interventional pulmonology technology. And about 10ml peripheral blood will be collected at the same time. The tissue will be sent to Pathology Department of Shanghai Chest Hospital and will be processed with paraffin-embedded, and for those diagnosed with nonsquamous NSCLC, the rest tissue will be extracted with DNA and performed NGS for the qualified DNA sample using Illumina Nextseq500 sequencer.The matched peripheral blood will also be extract with DNA and performed NGS using Illumina Nextseq500 sequencer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are suspected with nonsquamous non-small cell lung cancer according to the clinical, lab examination and imaging data and had never been diagnosed as primary lung cancer before will be enrolled into the study.
2. The clinical stage of the patients should be in stage IIIA-IV judged by the imaging data and can't receive surgery initially,
3. There exist at least one primary tumor and at least one enlarged LN which can be biopsied by minimally invasive techniques.

Exclusion Criteria:

1. The patient is highly suspected to benign lesion, small cell lung cancer and squamous cell carcinoma according to the clinical data.
2. Surgery was considered to be the primary treatment.
3. Patients who are diagnosed with lung cancer and received treatment with drugs or recurrent with lung cancer will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Gene mutations in matched samples | Up to one and a half years
  Gene mutations in primary tumor, matched metastatic LN and peripheral blood samples will be tested using NGS technique.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang S, Wang Z. Meta-analysis of epidermal growth factor receptor and KRAS gene status between primary and corresponding metastatic tumours of non-small cell lung cancer. Clin Oncol (R Coll Radiol). 2015 Jan;27(1):30-9. doi: 10.1016/j.clon.2014.09.014. Epub 2014 Oct 14. PMID 25445553
- [Background] Sherwood J, Dearden S, Ratcliffe M, Walker J. Mutation status concordance between primary lesions and metastatic sites of advanced non-small-cell lung cancer and the impact of mutation testing methodologies: a literature review. J Exp Clin Cancer Res. 2015 Sep 4;34(1):92. doi: 10.1186/s13046-015-0207-9. PMID 26338018
- [Background] Masago K, Fujita S, Muraki M, Hata A, Okuda C, Otsuka K, Kaji R, Takeshita J, Kato R, Katakami N, Hirata Y. Next-generation sequencing of tyrosine kinase inhibitor-resistant non-small-cell lung cancers in patients harboring epidermal growth factor-activating mutations. BMC Cancer. 2015 Nov 16;15:908. doi: 10.1186/s12885-015-1925-2. PMID 26572169
- [Background] Park S, Holmes-Tisch AJ, Cho EY, Shim YM, Kim J, Kim HS, Lee J, Park YH, Ahn JS, Park K, Janne PA, Ahn MJ. Discordance of molecular biomarkers associated with epidermal growth factor receptor pathway between primary tumors and lymph node metastasis in non-small cell lung cancer. J Thorac Oncol. 2009 Jul;4(7):809-15. doi: 10.1097/JTO.0b013e3181a94af4. PMID 19487967
- [Background] Gomez-Roca C, Raynaud CM, Penault-Llorca F, Mercier O, Commo F, Morat L, Sabatier L, Dartevelle P, Taranchon E, Besse B, Validire P, Italiano A, Soria JC. Differential expression of biomarkers in primary non-small cell lung cancer and metastatic sites. J Thorac Oncol. 2009 Oct;4(10):1212-20. doi: 10.1097/JTO.0b013e3181b44321. PMID 19687761
- [Background] Metzker ML. Sequencing technologies - the next generation. Nat Rev Genet. 2010 Jan;11(1):31-46. doi: 10.1038/nrg2626. Epub 2009 Dec 8. PMID 19997069